CLINICAL TRIAL: NCT06450093
Title: Comparative Clinical Evaluation of BioFlx, Zirconia, and Stainless-Steel Crowns in Primary Molars: A Randomized Controlled Clinical Trial
Brief Title: Comparative Clinical Evaluation of BioFlx, Zirconia, and Stainless-Steel Crowns in Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Elbadry, Assistant lecturer, peadiatric dentistry department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A0103024PP
Record Dates: First submitted 2024-06-02; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Dental Restoration
Keywords: Bioflx Crowns; Wear; Zirconia Crowns; stainless steel Crowns; periodontal changes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I Stainless steel crowns (control group) (Other): It will include 17 molars that will be restored by a stainless steel crown.
  Interventions: Other: Preformed stainless steel crown.
- Group II: Preformed zirconia crown (study group) (Other): It will include 17 molars that will be restored by Zirconia crowns.
  Interventions: Other: Preformed zirconia crown
- Group III: Preformed BioFlx crown (study group) (Other): It will include 17 molars that will be restored by BioFlx crowns.
  Interventions: Other: Preformed BioFlx crown

INTERVENTIONS:
Other: Preformed stainless steel crown. — A well-fitted preformed stainless-steel crown will be chosen by measuring the mesiodistal dimension of the tooth or its contralateral counterpart, using a graduated periodontal probe for guidance. (6) Tooth preparation will be carried out with #835 diamond fissure bur to reduce occlusal surface up to 1 to 1.5 mm. The interproximal reduction will be made mesially and distally using #169 L tapered diamond bur around 0.5 mm to clear the contact area creating a feather edge finish line. The selected crown size will be checked, and a trial fit will be done before cementation. The crown will be cemented using self-cured RMGI luting cement. The excess will be removed, and proper occlusion will be checked.
  Arms: Group I Stainless steel crowns (control group)
Other: Preformed zirconia crown — The material for crown restoration for this group is the preformed zirconia crown. Tooth preparation will be started by occlusal reduction (1 to 1.5 mm) using #835 diamond fissure bur. The interproximal reduction will be done mesially and distally with #169 L tapered diamond bur in such a way that a straight probe passes freely through the contact area. Rounding of line angles will be done and a knife-edge finish margin of the proximal surface will be obtained avoiding any ledge formation. The selected crown will be placed and checked for a passive fit. Consistent firm finger pressure will be applied during cementation with self-cured RMGI luting cement. Finally, crown placement will be checked.
  Arms: Group II: Preformed zirconia crown (study group)
Other: Preformed BioFlx crown — The prefabricated BioFlx crown will be used in this group. A similar-sized preformed crown will be selected. Tooth preparation will be carried out similarly to traditional SSCs with #835 diamond fissure bur for occlusal reduction by 1-1.5 mm including the central groove. The proximal preparation will be done mesially and distally with #169 L tapered diamond bur around 0.5 mm to clear the contact area creating a feather edge finish line. Placement of the crown will be achieved by a snug fit. Crown cementation will be carried out using self-cured RMGI luting cement and the excess cement will be removed using a floss or an explorer. (13) Finally, crown placement will be checked
  Arms: Group III: Preformed BioFlx crown (study group)

SUMMARY:
This study will be conducted to:

Evaluate and compare the clinical success, periodontal changes, and wear of antagonist teeth for three types of prefabricated crowns in primary molars: BioFlx crowns, Zirconia crowns, and Stainless Steel crowns.

DETAILED DESCRIPTION:
A randomized controlled clinical trial with three parallel groups, will be set up and reported according to the revised Consolidated Standards of Reporting Trials statement. The study will be conducted on 51 children with 51 molars aged between 4 and 7 years with a lower primary molar indicated for crown restoration. The children will be selected from the Pediatric Dental Clinic, Faculty of Dentistry, Mansoura University. They will be randomly divided into three equal groups (17 molars/each). Sequence generation and concealment will be done by a biostatistician who is not involved in the study. Group I (control group) will include stainless steel crowns, group II (study group) will include Zirconia crowns, group III (study group) will include BioFlx crowns. After obtaining the written consent form from the parents or guardians, the children will be randomly enrolled, and teeth will be assigned to the groups to receive the selected crowns. Clinical evaluation will be done concerning crown retention, color stability, secondary caries, periodontal changes, and wear of the opposing natural enamel. All crowns will be evaluated at the 3rd, 6th, 12th, and 18th months.

ELIGIBILITY:
Inclusion Criteria:

* Children who are free from any systemic disease.
* Children with a carious lower primary molar indicated for crown restoration.
* Teeth with an intact antagonist and neighboring primary molar.
* Cooperative children with scores 1 and 2 (positive or definitely positive) according to Frankl's behavior rating scale.

Exclusion Criteria:

* Children with extremely poor oral hygiene.
* Teeth showing radiographical furcation involvement or root resorption.
* Children with para-functional habits, bruxism, or deep bite.
* Teeth with inadequate non-restorable crown structure.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-10-04 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Crown retention | After 3, 6,12,18 months
  The crown retention will be measured concerning the proper adaptation of the crown or the complete crown loss according to the following:
  0 = present.
  1 = absent.
Color stability | After 3, 6,12,18 months
  The color stability will be evaluated using one crown from the original kit as a standard that will be held up to each crown restoration for color comparison according to the following:
  0= Unchanged.
  1= Minor deviation from original. 2 = Unacceptable discoloration.
Secondary caries | After 3, 6, 12,18 months
  Secondary caries will be measured according to USPHS by visual inspection with an explorer to inspect if there is evidence of caries with the margin of the crown restoration according to the following:
  0 = no caries
  1 = caries present
Gingival Index (Periodontal Changes) | After 3, 6, 12 ,18 months
  The GI (Gingival index) will be measured by the William Gingival Probe; the values will be recorded according to the following:
  0 = normal gingiva
  1. = mild inflammation: a slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation: redness, edema, glazing, or bleeding on probing
  3. = severe inflammation: marked redness or edema, a tendency toward spontaneous bleeding, and ulceration.
Periodontal Index (Periodontal changes) | After 3, 6, 12 ,18 months
  The PI (Periodontal Index) will be measured by the William Gingival probe; the values will be recorded according to the following:
  0 = no plaque
  1= film at the gingival margin and adjacent tooth 2 = moderate accumulation of plaque 3 = abundance of plaque.
Periodontal pocket depth (Periodontal changes) | After 3, 6, 12 ,18 months
  The PPD will be measured using a manual periodontal probe (UNC. 15 mm) according to the following:
  The pocket depth will be measured in mesiobuccal, distobuccal, mesiolingual, and distolingual areas. The periodontal probe will be inserted into the gingival sulcus parallel to the longitudinal axis of the tooth and then move in a walking fashion.
Wear of the opposing natural enamel. | After 12 months
  To evaluate the wear of the antagonistic natural enamel of the primary molar, alginate impressions will be taken immediately (baseline) and 1 year after cementation of the crowns. The resulting casts will be scanned using a 3D scanner and 3D software that will be used to calculate the maximum amount of linear wear using image superimposition techniques. The occlusal points of the crowns will be recorded in the software for measurements and comparisons, then it will be transformed into Standard Tessellation Language (STL) file format by the software

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University., Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No